CLINICAL TRIAL: NCT00003435
Title: A Pilot Study Involving Administration of Combination Anti-Retroviral Therapy and Transplantation of HLA-Matched Sibling Peripheral Blood Stem Cells or Partially HLA-Matched Unrelated Umbilical Cord Blood In Adults With HIV Infection and Hematologic Malignancies
Brief Title: Antiviral Therapy Plus Either Peripheral Stem Cell or Umbilical Cord Blood Transplantation in Treating Patients Who Are HIV Positive and Have Hematologic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066461; DUMC-97028; NCI-G98-1458
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2000-12

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult acute lymphoblastic leukemia; secondary acute myeloid leukemia; AIDS-related peripheral/systemic lymphoma; HIV-associated Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Antilymphocyte Serum; Melphalan; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: melphalan
Procedure: antiviral therapy
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Antiviral agents are drugs that act against viruses and may be an effective treatment for HIV. Peripheral stem cell transplantation or umbilical cord blood transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill tumor cells. Combining either umbilical cord blood transplantation or peripheral stem cell transplantation with antiviral therapy may be an effective treatment for HIV-positive patients who have hematologic cancer.

PURPOSE: Phase I trial to study the effectiveness of antiviral therapy plus either peripheral stem cell transplantation or umbilical cord blood transplantation in treating HIV-positive patients who have refractory or recurrent hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and safety of combination antiretroviral therapy followed by HLA matched sibling peripheral blood stem cell or unrelated umbilical cord blood transplants in HIV infected adults with hematologic malignancies. II. Measure the effects of this treatment on HIV viral burden in the serum and tissues of these patients. III. Measure immune reconstitution following treatment in this patient population.

OUTLINE: Patients receive a combination of 3 antiretroviral agents beginning at least 3 weeks prior to the initiation of the myeloablative conditioning regimen. The antiretroviral agents are discontinued on days -5 to -1 prior to transplant. Beginning on day 0 the antiretroviral agents are restarted and continue indefinitely. Patients who are given umbilical cord blood (UCB) transplants undergo collection of autologous peripheral blood stem cells (PBSC) prior to the myeloablative conditioning regimen in case there is UCB graft failure. Prior to PBSC or UCB transplantation on day 0, all patients receive a myeloablative conditioning regimen. The conditioning regimen consists of total body irradiation twice a day on days -9 to -5 and melphalan IV over 60 minutes on days -4 to -2. Patients receiving UCB transplant also receive anti-thymocyte globulin over 6 hours on days -3 to -1. Patients are followed every 3 months for 3 years, then annually for the next 3 years.

PROJECTED ACCRUAL: A total of 6 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed intermediate or high grade non-Hodgkin's lymphoma, acute myelogenous leukemia, or acute lymphocytic leukemia that is refractory to or relapsed after prior therapy Must be HIV seropositive confirmed by Western blot Must have a 6/6 HLA matched sibling donor or 6/6, 5/6, or 4/6 HLA matched umbilical cord blood (UCB) from the New York Blood Center's Unrelated UCB Bank that is not homozygous for the CCR-5 mutation No active primary CNS lymphoma or chronic CNS infection No history of AIDS defining opportunistic infection or active invasive aspergillus infection A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 to 55 Performance status: Karnofsky 70-100% Life expectancy: At least 6 months (unless due to hematologic malignancy) Hematopoietic: Peripheral CD4 count greater than 100/mm3 Hepatic: Transaminases no greater than 4 times normal Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction within the past 6 months Normal cardiac function (LVEF greater than 40%) Pulmonary: FVC and FEV1 greater than 70% of predicted DLCO at least 60% of predicted Other: No other malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix within the past 5 years Not pregnant (must have negative pregnancy test within 2 weeks of therapy)

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow, peripheral blood stem cell, or umbilical cord blood transplant Chemotherapy: Cumulative lifetime dose of doxorubicin no greater than 450 mg/m2 (or equivalent dose of mitoxantrone or daunorubicin) Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No concurrent involvement in any other clinical trial that may affect hematologic engraftment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Smith, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States